CLINICAL TRIAL: NCT03435861
Title: Effect of Neflamapimod (VX-745) on Brain Inflammation Using Positron Emission Tomography (PET) Scan in Alzheimer's Disease (AD) Patients
Brief Title: Effect of Neflamapimod on Brain Inflammation in Alzheimer's Disease Patients
Acronym: VIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Fondation Plan Alzheimer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC31/16/8371
Record Dates: First submitted 2017-12-22; First posted 2018-02-19 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — VX-745

STUDY DESIGN:
Intervention Model Description: Our mono-centric project will consist in a double-blinded randomized placebo-controlled study, assessing the effect of neflamapimod on brain inflammation in patients suffering of AD by using [18F]-DPA714
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VX-745 (Experimental): In the present study, VX-745 will be given at the dosage of 40 mg twice a day (1 tab. of 40 mg, twice), orally for 12 weeks
  Interventions: Drug: VX-745
- placebo (Placebo Comparator): In the present study, placebo will be given twice a day (1 tab. , twice), orally for 12 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: VX-745 — active drug capsules
  Other Names: neflamapimod
  Arms: VX-745
Drug: placebo — placebo capsules
  Arms: placebo

SUMMARY:
For this project, neflamapimod and placebo will be provided free of charge by the EIP company (www.eippharma.com). Neflamapimod is currently tested in 2 clinical trials in AD, one in Europe (The Netherlands) and one in the USA (clinical trials.gov/VX-745). The company commenced in May 2015 dosing in two phase 2a clinical studies in patients with Early AD: one in the Netherlands that is focused on PET amyloid imaging as the primary biomarker of drug effect, and one in the US (California) that is focused on Cerebrospinal fluid (CSF) evaluation to determine CSF drug concentrations and effects on inflammatory markers and disease biomarkers. Pharmacokinetic evaluation in these patients has demonstrated blood drug concentration levels in the predicted therapeutic range; and importantly, the data from the US study demonstrate that the drug achieves target drug concentrations in CSF, thus confirming the drug robustly enters the brain in humans.

The present project offers us a unique chance to test this promising drug in AD patients. The aim of the study is to focus on PET neuroinflammation imaging as the primary biomarker of this drug effect. The chosen biomarker for imaging neuroinflammation in patients is [1 8F]-DPA714.

DETAILED DESCRIPTION:
The present project is an intervention proof of concept study to test the efficacy of neflamapimod in a population of AD patients at an early stage.

To track the impact of this drug in patients, the investigators will use an innovative radiotracer, [18F]DPA-714, as a promising ligand of microglial activation targeting the translocator protein (TSPO), specific of microglial activation. The use of [18F]DPA-714 will allow to monitor the evolution of neuroinflammation in patients as a function of treatment. The main objective will be to compare the level of inflammation using the [18F]DPA-714 in neflamapimod and placebo groups after 12 weeks of treatment. Blood and cerebrospinal fluid (CSF) samples and magnetic resonance imaging (MRI) will also be collected to assess inflammation markers and brain structure respectively in these patients.

ELIGIBILITY:
Inclusion Criteria:

* A group of 40 AD patients at an early stage (prodromal) will be recruited. Patient's recruitment will follow the most recent research criteria for AD in its "typical form" (Dubois, Feldman et al. 2014):

  * Age 50 - 90 (inclusive)
  * Willing and able to provide informed consent
  * Objective memory impairment corroborated by level of performance on a standardized memory test (Free and Cued Selective Reminding test, (Grober, Hall et al. 2008)) < -1.5 DS according to established norms and
  * Documented cerebral amyloidopathy using CSF analysis or PET amyloid imaging and
  * Early stage of the disease (Mini Mental State Examination > 20) (Folstein, Robins et al. 1983).

Exclusion Criteria:

* • Evidence of neurodegenerative disease other than AD

  * Inability for any reason to undergo MRI scans (e.g. pacemaker). Patients who require sedation for screening procedures such as MRI may receive a short-acting sedative.
  * Psychiatric disorder that would compromise ability to comply with study requirements
  * History of cancer within the last 5 years, except basal cell carcinoma, non-squamous skin carcinoma, prostate cancer or carcinoma in situ with no significant progression over the past 2 years
  * Significant cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder or metabolic/endocrine disorders or other disease that would preclude treatment with p38 MAP kinase inhibitor and/or assessment of drug safety and efficacy
  * Recent (<60 days) changes to AD medications prescribed for cognitive reasons or with the potential to impact cognition
  * Psychotropic drugs taken within 1 month. Anticoagulant drugs taken within 1 week.
  * Participation in a study of an investigational drug less than 6 months or 5 half-lives of the investigational drug, whichever is longer, before enrollment in the study
  * Male subjects with female partner of child-bearing potential who are unwilling or unable to adhere to contraception requirements
  * Female subjects who have not reached menopause or have not had a hysterectomy or bilateral oophorectomy/salpingoophorectomy
  * Positive urine or serum pregnancy test or plans desires to become pregnant during the course of the trial
  * History of alcohol and/or illicit drug abuse within 6 months.
  * Infection with hepatitis A, B or C or HIV.
  * Any factor deemed by the investigator to be likely to interfere with study conduction

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
brain inflammation assessed by [18F]-DPA714, Standard Uptake Value (SUV) | 3 month
  To track the impact of this drug in patients, investigators will use an innovative radiotracer, [18F]DPA-714, as a promising ligand of microglial activation targeting the translocator protein (TSPO), specific of microglial activation. The use of [18F]DPA-714 will allow us to monitor the evolution of neuroinflammation in patients as a function of treatment. the main objective will be to compare the level of inflammation using the [18F]DPA-714 in neflamapimod and placebo.
  Regional cortical DPA-714 mean SUV will be measured in each subject using a Matlab (The MathWorks®) script. Mean global SUVs will be calculated
brain inflammation assessed by [18F]-DPA714, Standard Uptake Value (SUV) 2 | 3 month
  SUVs in the five lobes will be calculated.
brain inflammation assessed by [18F]-DPA714, Standard Uptake Value (SUV)3 | 3 month
  SUVs in specific regions of interest (ROIs: orbitofrontal, anterior cingulate, posterior cingulate and precuneus) will be calculated.

SECONDARY OUTCOMES:
Neuropsychological assessment to assess the following cognitive functions 1: | 3 month
  Memory: Rey Figure
Neuropsychological assessment to assess the following cognitive functions 2: | 3 month
  Memory: DMS 48,
Neuropsychological assessment to assess the following cognitive functions 1.1: | 3 month
  Language: confrontation naming (Gremots),
Neuropsychological assessment to assess the following cognitive functions 2.2: | 3 month
  Language: FAS fluencies,
Neuropsychological assessment to assess the following cognitive functions 3: | 3 month
  o Attention and executive functions: D2
Neuropsychological assessment to assess the following cognitive functions 4: | 3 month
  o Attention and executive functions: TEA
Neuropsychological assessment to assess the following cognitive functions 5: | 3 month
  o Attention and executive functions: SDMT WAIS
Blood and CSF biomarkers of inflammation1 | 3 month
  ApoE phenotype
Blood and CSF biomarkers of inflammation 2 | 3 month
  TSPO phenotype,
Blood and CSF biomarkers of inflammation 3 | 3 month
  TNFa,
Blood and CSF biomarkers of inflammation 4 | 3 month
  IL-1b,
Blood and CSF biomarkers of inflammation 5 | 3 month
  IFNg
Blood and CSF biomarkers of inflammation 6 | 3 month
  IL-12
Blood and CSF biomarkers of inflammation 7 | 3 month
  IFNa/b
Blood and CSF biomarkers of inflammation 8 | 3 month
  IL-10
Blood and CSF biomarkers of inflammation 9 | 3 month
  IL-6
Blood and CSF biomarkers of inflammation 10 | 3 month
  IL-8,
Blood and CSF biomarkers of inflammation 11 | 3 month
  MCP-1,
Blood and CSF biomarkers of inflammation 12 | 3 month
  GM-CSF
Blood and CSF biomarkers of inflammation 13 | 3 month
  IL-27
Blood and CSF biomarkers of inflammation 14 | 3 month
  chimiokines receptors,
Blood and CSF biomarkers of inflammation 15 | 3 month
  PD-1,
Blood and CSF biomarkers of inflammation 16 | 3 month
  CD14/16
Blood and CSF biomarkers of inflammation 17 | 3 month
  p-tau,
Blood and CSF biomarkers of inflammation 18 | 3 month
  abéta42,
Blood and CSF biomarkers of inflammation 19 | 3 month
  Abeta40,
Blood and CSF biomarkers of inflammation 20 | 3 month
  cells count
Blood and CSF biomarkers of inflammation 21 | 3 month
  TNFa
Blood and CSF biomarkers of inflammation 22 | 3 month
  IL-1b
Blood and CSF biomarkers of inflammation 23 | 3 month
  IL-12
Blood and CSF biomarkers of inflammation 24 | 3 month
  MCP-1
Blood and CSF biomarkers of inflammation 25 | 3 month
  GM-CSF
Blood and CSF biomarkers of inflammation 26 | 3 month
  IL-27,
Blood and CSF biomarkers of inflammation 27 | 3 month
  PD-1
Blood and CSF biomarkers of inflammation 28 | 3 month
  CD14/16

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie PARIENTE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tormahlen NM, Martorelli M, Kuhn A, Maier F, Guezguez J, Burnet M, Albrecht W, Laufer SA, Koch P. Design and Synthesis of Highly Selective Brain Penetrant p38alpha Mitogen-Activated Protein Kinase Inhibitors. J Med Chem. 2022 Jan 27;65(2):1225-1242. doi: 10.1021/acs.jmedchem.0c01773. Epub 2021 May 11. PMID 33974419